CLINICAL TRIAL: NCT02160808
Title: Secretin Infusion to Prevent Pancreatic Leaks Following Pancreatic Resection
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Timothy Gardner, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D13208 TBG-01
Record Dates: First submitted 2014-05-13; First posted 2014-06-11 (Estimated); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Injury of Body of Pancreas
MeSH Terms: interventions — Secretin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Secretin (Active Comparator): Stimulate pancreatic secretion
  Interventions: Drug: Secretin
- Saline (Placebo Comparator): Placebo should not stimulate the pancreas to release its fluids
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Secretin — Drug to stimulate pancreatic secretion
  Arms: Secretin
Drug: Placebo
  Arms: Saline

SUMMARY:
Pancreatic leaks complicate pancreatic resection in approximately 20% of cases. The pancreatic anastomosis or repair has been referred to as the Achilles heel of pancreatic surgery. Unfortunately, despite recognition of this problem and multiple operative techniques proposed to prevent this complication, leaks continue to represent a major cause of morbidity for patients undergoing pancreatic surgery. Treatment of leaks often requires nutritional support with total parenteral nutrition to diminish the leak in addition to invasive interventions to contain the leak with drains, stents or in severe cases, reoperation. Experiential data suggest that intra-operative infusions of secretin, a naturally occurring hormone that stimulates bicarbonate release from the pancreas, following resection but just prior to abdomen closure, may identify a leak if present. If secretin can demonstrate evidence of leaking intra-operatively, the pancreatic duct leak may be able to be fixed prior to abdominal closure. The investigators aim to determine if giving an intra-operative infusion of secretin will allow for identification and treatment of leaks after pancreatic reconstruction and prior to abdominal closure, leading to a reduction in the rate of pancreatic anastomotic leaks requiring intervention. The investigators will perform a double-blind, randomized pilot study of 176 patients undergoing pancreatic resection (pancreaticoduodenectomy and distal pancreatectomy) at Dartmouth-Hitchcock Medical Center. 88 of those patients will receive an intra-operative secretin infusion prior to abdominal closure and 88 will receive a saline placebo. Our primary outcome of interest will be the rate of pancreas duct leaks in each group as measured by the concentration of amylase present in the surgical drains 3 days following surgery.

DETAILED DESCRIPTION:
We hypothesize that intra-operative, intravenous secretin administration will decrease the rate of pancreatic leaks in patients undergoing pancreatic resection. Our primary objective is to determine if intravenous secretin administration will decrease the amount of pancreatic leaks as measured by the 2016 ISGPS definition of pancreatic leaks. Our 1) secondary objectives are to determine if intra-operative intravenous secretin administration changes the management of the pancreatic resection margin intra-operatively and 2) Length of hospital stay.

Use a level of detail similar to what would be used when submitting an article for publication in a peer reviewed journal. Explain the study procedures, data collection, and analysis process. Please define terms and explain concepts which might be confusing to reviewers who are not expert in the area of the study. If a formal protocol for the study exists, page references to the protocol are acceptable.

This study design is a prospective, double-blind, randomized-controlled trial. We will enroll patients in our institution undergoing pancreatic resection to receive either 1) one dose weight-based Secretin to be given once the closure of the pancreatic resection margin is complete 2) saline placebo.

Consent and basic demographics will be garnered by the physician in an office visit once the surgery has been scheduled and consent for the surgery is being obtained. The consent will be validated by the treating surgeon in the pre-procedure area on the day of the surgery.

The patient will undergo the scheduled surgery. Once the pancreatic anastomosis has been deemed acceptable by the attending physician, but prior to abdominal closure, the patient will be randomized to receive either Secretin (0.2 mcg/kg) or saline placebo. The attending surgeon will be blinded to this assignment.

10 minutes after receiving the Secretin or placebo, the attending surgeon will examine the anastomosis or repaired cut edge of the pancreas to determine if leakage of pancreatic fluid is noted, leak location(s), type (side branch/main duct) and whether any further intervention was performed in an effort to close the leak. Specifics of operative intervention will be documented. The patient will then undergo standard surgical closure of the abdomen.

As is standard of care at DHMC, surgical drains will be placed adjacent to the anastomosis and drain amylase output will be checked on POD #1, POD#3 and POD#5. Pancreatic leak is defined according to the International Study Group of Pancreatic Fistula (ISGPF) definition as amylase drainage of greater than a 3-fold elevation above the upper limit of normal in serum through the surgically placed drains on POD #3. Randomization assignments will be revealed once the patient has been discharged from the hospital following their initial surgical intervention. A follow-up visit with the patient two weeks following discharge, will evaluate for any evidence of ongoing pancreatic duct leak.

The primary outcome of interest will be the presence of pancreatic leaks based on the drain amylase on POD#3. Secondary outcomes will include the technical interventions intra-operatively directed to leak closure or manipulation of the anastomosis following Secretin or placebo stimulation and the length of hospitalization.

Patient demographics, risk factors, operative technique, randomization assignment and outcome data will be recorded on standard case report forms - See Case Report Forms in Appendix. Data will be stored in an encrypted hard-drive by a single agent (Gardner) who is the only researcher who has access to the randomization data.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled for pancreatic surgery requiring pancreatic resection at DHMC
2. Age greater than 18 years old
3. Ability to provide written informed consent

Exclusion Criteria:

1. Inability to provide written informed consent
2. Current ongoing acute pancreatitis
3. Pregnant or nursing mothers
4. Any medical condition which in the judgment of the Investigator renders participation in this study medically inadvisable.
5. Participation in an investigational clinical study for a drug or medical device within 30 days prior to Visit 1.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-09-21 (Actual); Study Completion 2019-09-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Smith KD, Barth RJ, Colacchio TA, Chevalier JI, Bergmann LE, Purich ED, Gardner TB. Effect of intraoperative secretin on operative outcomes in pancreatic resection: A randomized controlled trial. Pancreatology. 2021 Apr;21(3):515-521. doi: 10.1016/j.pan.2021.02.002. Epub 2021 Feb 8. PMID 33602643

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline: Placebo should not stimulate the pancreas to release its fluids
  Placebo
Period: Overall Study
Arm/Group | Secretin | Saline
Started | 87 | 83
Completed | 87 | 83
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secretin | Saline | Total
Number analyzed (Participants) | 87 | 83 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (12.3) | 63.5 (12.1) | 63.45 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 33 | 76
  Male | 44 | 50 | 94
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.6 (5.0) | 26.7 (6.3) | 26.65 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biochemical Leak/Grade B Fistula/Grade C Fistula
Description: Outcome based on revised ISGPS Guidelines which require a three day drain amylase concentration greater than 3x the normal serum amylase concentration. Biochemical leaks are the mildest for of fistula which have no clinical consequence. Grade B fistula are more severe requiring usually percutaneous drainage placement. Grade C fistula are most severe resulting in significant morbidity and/or death.
Time Frame: 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Secretin | Saline
Number analyzed (Participants) | 87 | 83
Participants
  Biochemical Leak | 25 | 16
  Grade B Fistula | 3 | 5
  Grade C Fistula | 0 | 0

2. Secondary Outcome: Number of Participants With Intra-operative Intervention, Subsequent Biochemical Leak or B/C Fistula After Drug Administration
Description: Following the administration of Secretin or Placebo intraoperatively, the surgeon will have the opportunity to evaluate the anastomosis to determine if there is ongoing leak. If there is ongoing leak, then the surgeon will be able to treat the leak intra-operatively prior to operative closure. In those patients in whom an intervention was performed, they were subsequently evaluated to determine if they developed a biochemical leak or grade B/C fistula.
Time Frame: Through completion of intra-operative intervention and subsequent biochemical leak, B/C Fistula up to 30 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Secretin | Saline
Number analyzed (Participants) | 87 | 83
Participants
  Intervention | 8 | 3
  Subsequent Biochemical Leak | 8 | 2
  Subsequent B/C Fistula | 0 | 1

3. Secondary Outcome: Length of Hospitalization
Description: Surrogate marker for operative success
Time Frame: Duration of study - average 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Secretin | Saline
Number analyzed (Participants) | 87 | 83
Days | 10.3 (6.5) | 10.2 (5.5)

ADVERSE EVENTS:
Time Frame: Study enrollment until 30 days post-hospital discharge, an average of 45 days
Arm/Group | Secretin | Saline
All-Cause Mortality (participants affected / at risk) | 0/87 | 1/83
Serious Adverse Events (participants affected / at risk) | 15/87 | 32/83
Other Adverse Events (participants affected / at risk) | 36/87 | 23/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secretin (N=87) | Saline (N=83)
Bile Leak (Hepatobiliary disorders) | 1 | 3
Deep Surgical Site Infection (Surgical and medical procedures) | 3 | 3
Gastroparesis (Gastrointestinal disorders) | 0 | 1
Hemorrhage (Surgical and medical procedures) | 6 | 10
Hernia (Surgical and medical procedures) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 2
Infection - other (Infections and infestations) | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 2
Superficial surgical site infection (Infections and infestations) | 1 | 6
Other (Surgical and medical procedures) | 3 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secretin (N=87) | Saline (N=83)
Chyle Leak (Hepatobiliary disorders) | 3 | 1
Deep Surgical Site Infection (Surgical and medical procedures) | 1 | 0
Gastroparesis (Gastrointestinal disorders) | 2 | 1
Hemorrhage (Surgical and medical procedures) | 3 | 5
Hernia (Surgical and medical procedures) | 0 | 1
Hypertension (Cardiac disorders) | 7 | 2
Hypotension (Cardiac disorders) | 10 | 5
Infection - other (Infections and infestations) | 1 | 3
Superficial Surgical Site Infection (Surgical and medical procedures) | 6 | 4
Other (Surgical and medical procedures) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT02160808/Prot_SAP_000.pdf